CLINICAL TRIAL: NCT02462928
Title: Safety and Efficacy of Abicipar Pegol (AGN-150998) in Patients With Neovascular Age-related Macular Degeneration (CEDAR Study)
Brief Title: A Safety and Efficacy Study of Abicipar Pegol in Participants With Neovascular Age-related Macular Degeneration
Acronym: CEDAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 150998-005; 2014-004579-22 (EudraCT Number); CEDAR (Other: Allergan)
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Results first posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — abicipar pegol; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Abicipar Pegol 2 mg (2Q8) (Experimental): Abicipar pegol 2 mg was administered to the study eye by intravitreal injection on Day 1, Week 4, Week 8 and every 8 weeks (2Q8) thereafter through Week 96. Scheduled visits occurred every 4 weeks. To maintain masking, sham was administered to the study eye at scheduled visits where abicipar was not administered.
  Interventions: Drug: Abicipar Pegol; Other: Sham Procedure
- Abicipar Pegol 2 mg (2Q12) (Experimental): Abicipar pegol 2 mg was administered to the study eye by intravitreal injection on Day 1, Week 4, Week 12, and every 12 weeks (2Q12) thereafter through week 96. Scheduled visits occurred every 4 weeks. To maintain masking, sham was administered to the study eye at scheduled visits where abicipar was not administered.
  Interventions: Drug: Abicipar Pegol; Other: Sham Procedure
- Ranibizumab 0.5 mg (rQ4) (Active Comparator): Ranibizumab (Lucentis®) 0.5 mg was administered to the study eye by intravitreal injection every 4 weeks (rQ4) from Day 1 through Week 96.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Abicipar Pegol — Abicipar pegol intravitreal injection.
  Other Names: AGN-150998
  Arms: Abicipar Pegol 2 mg (2Q12); Abicipar Pegol 2 mg (2Q8)
Drug: Ranibizumab — Ranibizumab intravitreal injection.
  Other Names: Lucentis®
  Arms: Ranibizumab 0.5 mg (rQ4)
Other: Sham Procedure — Sham injection.
  Arms: Abicipar Pegol 2 mg (2Q12); Abicipar Pegol 2 mg (2Q8)

SUMMARY:
This is a safety and efficacy study of abicipar pegol in participants with neovascular age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of age-related macular degeneration in at least 1 eye
* Best corrected visual acuity of 20/40 to 20/320 in the study eye
* Best corrected visual acuity of 20/200 or better in the non-study eye

Exclusion Criteria:

* History of vitrectomy, macular surgery, or glaucoma surgery in the study eye
* Cataract or refractive surgery in the study eye within the last 3 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 939 (Actual)
Dates: Start 2015-06-25 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2019-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Li, Study Director — Allergan
Locations (151):
- United States (71):
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Associated Retina Consultants, Ltd., Phoenix, Arizona
  - Arizona Retina and Vitreous Consultants, Phoenix, Arizona
  - Retina Associates Southwest, P.C., Tucson, Arizona
  - The Retina Partners, Encino, California
  - Retina Consultants of Orange County, Fullerton, California
  - Mark B. Kislinger MD Inc., Glendora, California
  - Atlantis Retina Institute (Atlantis Eyecare), Huntington Beach, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Northern California Retina Vitreous Associates Medical Group, INC., Mountain View, California
  - Retina Institute of California, Palm Desert, California
  - Doheny Vision Research, Pasadena, California
  - Orange County Retina Medical Group, Santa Ana, California
  - California Retina Consultants, Santa Barbara, California
  - Retina Eye Specialists, South Pasadena, California
  - Colorado Retina Associates, Golden, Colorado
  - Retina Health Center, Fort Myers, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - Ocala Eye PA, Ocala, Florida
  - Magruder Eye Institute, Orlando, Florida
  - Retina Care Specialists, Palm Beach Gardens, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Retina Vitreous Associates of Florida - Saint Petersburg, St. Petersburg, Florida
  - USF Eye Institute, Tampa, Florida
  - Georgia Retina, P.C., Marietta, Georgia
  - Marietta Eye Clinic - Main Office, Marietta, Georgia
  - Thomas Eye Group, PC, Sandy Springs, Georgia
  - Retina Consultants of Hawaii, Inc., ‘Aiea, Hawaii
  - Gailey Eye Clinic, Bloomington, Illinois
  - Carle at the Fields, Champaign, Illinois
  - University Retina and Macula Associates, PC, Lemont, Illinois
  - Raj K. Maturi, MD, PC, Indianapolis, Indiana
  - John Kenyon American Eye Institute, New Albany, Indiana
  - Ochsner Health Center, New Orleans, Louisiana
  - Retina Specialists, Baltimore, Maryland
  - The Bert M Glaser National Retina Institute, Towson, Maryland
  - Lahey Medical Center, Peabody, Massachusetts
  - Kellog Eye Center - University of Michigan Health System, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Sierra Eye Associates, Reno, Nevada
  - Retina Associates of New Jersey, Teaneck, New Jersey
  - Capital Region Retina, PLLC, Albany, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Long Island Vitreoretinal Consultants, Great Neck, New York
  - Ophthalmic Consultants of Long Island, Oceanside, New York
  - Retina Associates of Western New York, Rochester, New York
  - Island Retina, Shirley, New York
  - Carolina Eye Associates, Southern Pines, North Carolina
  - Wake Forest Baptist Health Eye Center, Winston-Salem, North Carolina
  - Apex Eye Clinical Research, Fairfield, Ohio
  - Lancaster Retina Specialists, Lancaster, Pennsylvania
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Associates in Ophthalmology, Ltd., West Mifflin, Pennsylvania
  - Retina Consultants of Carolina, Greenville, South Carolina
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Retina Research Institute of Texas, Abilene, Texas
  - Texas Retina Associates, Arlington, Texas
  - Texan Eye, Austin, Texas
  - TX Retina Associates, Dallas, Texas
  - Houston Eye Associates (HEA) - Gramercy Location, Houston, Texas
  - Retina and Vitreous of Texas, Houston, Texas
  - Retinal Consultants of Houston, Houston, Texas
  - San Antonio Eye Center, San Antonio, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - Retina Associates of Utah, Salt Lake City, Utah
  - University of Virginia - Department of Ophthalmology, Charlottesville, Virginia
  - Piedmont Eye Center, Inc., Lynchburg, Virginia
  - Retina Institute of Virginia, Richmond, Virginia
- Argentina (9):
  - Clinica Privada Kaufer Cataract Center, Martínez, Buenos Aires
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Centro Oftalmologico Rosario SRL, Rosario, Santa Fe Province
  - Grupo Laser Vision, Rosario, Santa Fe Province
  - Organizacion Medica de Investigacion, Buenos Aires
  - Instituto Oftalmologico de Buenos Aires - Oftalmos, Buenos Aires
  - Centro Privado de Ojos Romagosa, Córdoba
  - Instituto Oftalmologico de Cordoba, Córdoba
  - Oftar Centro Privado de Oftalmologia, Mendoza
- Austria (4):
  - Medical University Graz, Graz
  - Medizinische Universitat Innsbruck, Univ., Innsbruck
  - Kepler Universitatsklinikum GmBH, Linz
  - Konventhospital Barmherzige Brueder Linz, Linz
- Chile (2):
  - KYDOFT, Santiago, Las Condes
  - Instituto Oftalmologica Profesor Arentsen, Santiago, Santiago Metropolitan
- Colombia (2):
  - Centro Medico Imbanaco, Cali, Valle del Cauca Department
  - Fundacion Oftalmologica Nacional - FUNDONAL, Bogotá
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Kralovske Vinohrady Oftalmologicka klinika, Prague
  - Vseobecna fakultni nemocnice v Praze Ocni Klinika, Prague
- France (6):
  - Hopital Pellegrin, Bordeaux
  - Centre Hospitalier Intercommunal de Creteil, Créteil
  - Hopital de la Croix Rousse, Service d'Opthalmologie, Lyon
  - CHU de Nantes, Nantes
  - Centre Ophtalmologique d'Imagerie et de Laser, Paris
  - Centre Ophtalmologique Saint Exupery, Saint-Cyr-sur-Loire
- Germany (10):
  - Dardenne Eye Hospital, Bad Godesberg
  - Klinikum Dresden Friedrichstadt, Dresden
  - Internationale Innovative Ophthalmochirurgie Breyer & Kaymak & Klabe Augenchirurgie, Düsseldorf
  - Eye Center, University of Freiburg, Freiburg im Breisgau
  - Universitats-augenklinik Gottingen, Göttingen
  - Stadtisches Klinikum, Karlsruhe
  - Universitätsklinikum Leipzig AöR Klinik und Poliklinik für Augenheilkunde, Leipzig
  - Universitätsklinikum Giessen und Marburg GmbH, Marburg
  - Augenklinik im Dietrich-Bonhoeffer - Klinikum Neubrandenburg, Neubrandenburg
  - Clinic and policlinic of ophthalmology, University of Regensburg, Regensburg
- Hong Kong (2):
  - The University of Hong Kong, Aberdeen
  - The Chinese University of Hong Kong Hongkong eye hospital, Kowloon
- Israel (10):
  - Bnai Zion Medical Center (BZMC) Technion-Israel Institute of Technology, Haifa
  - Rambam Health Care Campus, Haifa
  - Carmel Medical Center Ophthalmology Clinic, Haifa
  - Edith Wolfson Medical Center, Holon
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center Beilinson Hospital, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - TASMC (The Tel-Aviv Sourasky Medical Centre), Tel Aviv
  - Chaim Sheba Medical Center Goldschleger Eye Clinic Sheba Medical Center, Tel Litwinsky
  - Shamir Medical Centre, Ẕerifin
- Pauls Stradins Clinical University Hospital Opthalmology Clinic, Riga, LV, Latvia
- New Zealand (2):
  - Auckland Eye, Remuera, Auckland
  - University of Auckland, Auckland
- Philippines (5):
  - Cebu Doctors University Hospital, Cebu City, National Capital Region
  - Asian Eye Institute, Makati City, National Capital Region
  - Pacific Eyecare and Laser Institute, Makati City, National Capital Region
  - The Medical City, Pasig, National Capital Region
  - St. Luke's Medical Center, Quezon City, National Capital Region
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore National Eye Centre- Singapore Eye Research Institute (SNECSERI), Singapore
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic Univ. Of Seoul St. Mary's Hospital, Seocho, Seoul
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System Serverance Hospital, Seoul
- Spain (13):
  - Centro de Oftalmologia Barraquer, Barcelona
  - Institut Clinic d'Oftalmologia Hospital Clinic de Barcelona, Barcelona
  - Instituto de Microcirugía Ocular DOS, S.L.U Area de Consultas, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Valles Oftalmologia Research Hospital, Barcelona
  - Instituto Clínico Quirúrgico de Oftalmología (ICQO), Bilbao
  - Hospital Clinico San Carlos, Madrid
  - Clinica Universidad de Navarra Servicio de Oftalmologia, Pamplona
  - Hospital General de Valencia Unidad de Investigacion Clinica, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Clinico Universitario, Valladolid
  - Hospital Clínico Universitario Lozano Blesa. Unidad de Retina Médica y Quirúrgica, Zaragoza
  - Hospital Miguel Servet, Zaragoza
- Switzerland (3):
  - Universitatsklinik fur Augenheilkunde, Inselspital, Bern
  - VISTA Klinik Binningen, Binningen
  - Stiftung für wissenschaftliche Forschung am Stadtspital Triemli, Zurich

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abicipar Pegol 2 mg (2Q8) | Abicipar Pegol 2 mg (2Q12) | Ranibizumab 0.5 mg (rQ4)
Started | 314 | 313 | 312
Completed | 224 | 221 | 255
Not Completed | 90 | 92 | 57
Not completed — Screen Failure:Missed Exclusion Criteria | 1 | 1 | 2
Not completed — Adverse Event | 47 | 51 | 25
Not completed — Lack of Efficacy | 3 | 8 | 3
Not completed — Lost to Follow-up | 4 | 4 | 1
Not completed — Withdrawal by Patient | 31 | 21 | 21
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Reason not Specified | 4 | 6 | 5

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Abicipar Pegol 2 mg (2Q8) | Abicipar Pegol 2 mg (2Q12) | Ranibizumab 0.5 mg (rQ4) | Total
Number analyzed (Participants) | 314 | 313 | 312 | 939
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.5 (8.4) | 76.9 (8.0) | 77.1 (8.4) | 76.5 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 183 | 169 | 514
  Male | 152 | 130 | 143 | 425
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 249 | 248 | 243 | 740
  Black | 2 | 1 | 1 | 4
  Asian | 49 | 44 | 45 | 138
  Hispanic | 12 | 12 | 11 | 35
  Not Reported | 2 | 8 | 12 | 22
Best-corrected Visual Acuity (BCVA) Per Per-protocol Population [Mean (Standard Deviation); unit: letters] — BCVA was measured using eye chart and reported as number of letters read correctly using the ETDRS Scale (ranging from 0 to 100 letters) in study eye. Lower number of letters read correctly on eye chart, worse the vision (or visual acuity). Study eye is defined as eye that meets entry criteria. If both eyes met entry criteria, eye with worse BCVA at baseline (Day 1) was selected as study eye. If both eyes had same BCVA values at baseline (Day 1), then participant had to select their non-dominant eye for treatment, or else right eye was selected as study eye. Population: The per-protocol (PP) population included all randomized and treated participants without any protocol deviations that impacted the primary efficacy variable and with treatment compliance to represent the intended regimen adequately.
  letters
    number analyzed (Participants) | 265 | 262 | 290 | 817
    (all) | 56.7 (13.3) | 56.3 (13.1) | 56.5 (12.6) | 56.5 (13.0)
BCVA Per ITT Population [Mean (Standard Deviation); unit: letters] — BCVA was measured using eye chart and reported as number of letters read correctly using the ETDRS Scale (ranging from 0 to 100 letters) in study eye. Lower number of letters read correctly on eye chart, worse the vision (or visual acuity). Study eye is defined as eye that meets entry criteria. If both eyes met entry criteria, eye with worse BCVA at baseline (Day 1) was selected as study eye. If both eyes had same BCVA values at baseline (Day 1), then participant had to select their non-dominant eye for treatment, or else right eye was selected as study eye. Population: Number analyzed is the number of participants with data available at Baseline.
  letters
    number analyzed (Participants) | 313 | 313 | 312 | 938
    (all) | 56.4 (13.4) | 56.5 (12.9) | 56.5 (12.5) | 56.5 (12.9)
Central Retinal Thickness (CRT) [Mean (Standard Deviation); unit: microns] — CRT was assessed using spectral domain optical coherence tomography (SD-OCT), a non-invasive diagnostic system providing high-resolution imaging sections of the retina. SD-OCT was performed in the study eye after pupil dilation. The study eye is defined as the eye that meets the entry criteria. If both eyes met the entry criteria, the eye with the worse BCVA at baseline (Day 1) was selected as the study eye. If both eyes had same BCVA values at baseline (Day 1), then the participant had to select their non-dominant eye for treatment, or else the right eye was selected as the study eye. Population: Number analyzed is the number of participants with data available at Baseline.
  microns
    number analyzed (Participants) | 313 | 313 | 312 | 938
    (all) | 384.7 (142.7) | 378.4 (119.1) | 378.2 (120.5) | 380.4 (127.8)
National Eye Institute Visual Functioning Questionnaire-25 (NEI-VFQ-25) [Mean (Full Range); unit: score on a scale] — NEI-VFQ-25 consists of 25 vision-targeted questions that represent 11 vision-related quality of life subscales and one general health item. Responses of individual participants were recorded as scores that ranged between 0 (worst) to 100 (best vision related function) with higher scale indicating better vision related function. The overall composite score is then calculated by averaging over all 11 vision-targeted subscale scores, excluding the general health score. Overall composite score was calculated based on mean of non-missing subscales. Population: Number analyzed is the number of participants with data available at Baseline.
  score on a scale
    number analyzed (Participants) | 313 | 313 | 311 | 937
    (all) | 78.7 [28 to 98] | 77.3 [34 to 98] | 77.1 [23 to 100] | 77.7 [23 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Stable Vision at Week 52
Description: Stable vision was defined as a loss of fewer than 15 letters in BCVA compared to baseline. BCVA was measured using an eye chart and reported as the number of letters read correctly using the Early Treatment of Diabetic Retinopathy Study (ETDRS) Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. The percentage of participants with a BCVA loss of fewer than 15 letters are reported. The study eye is defined as the eye that meets the entry criteria. If both eyes met the entry criteria, the eye with the worse BCVA at baseline (Day 1) was selected as the study eye. If both eyes had same BCVA values at baseline (Day 1), then the participant had to select their non-dominant eye for treatment, or else the right eye was selected as the study eye.
Time Frame: Baseline to Week 52
Population: The per-protocol (PP) population included all randomized and treated participants without any protocol deviations that impacted the primary efficacy variable and with treatment compliance to represent the intended regimen adequately.
Measure: Number; unit: percentage of participants
Arm/Group | Abicipar Pegol 2 mg (2Q8) | Abicipar Pegol 2 mg (2Q12) | Ranibizumab 0.5 mg (rQ4)
Number analyzed (Participants) | 265 | 262 | 290
percentage of participants | 91.7 | 91.2 | 95.5
Statistical Analysis 1: Comparison: Abicipar Pegol 2 mg (2Q8) vs Ranibizumab 0.5 mg (rQ4); Test type: Non-Inferiority — For hypothesis testing, if the lower limit of 95.1% Confidence Interval (CI) for the difference between an abicipar group and ranibizumab was greater than or equal to -10%, non-inferiority of abicipar was established; Percentage Difference = -3.8, 95.1% CI 2-sided [-8.2 to 0.3] — The 95.1% CI for the weighted difference were calculated based on the Newcombe method using the Cochran-Mantel-Haenszel weights and baseline BCVA (≤55 vs >55 letters) as stratification factor
Statistical Analysis 2: Comparison: Abicipar Pegol 2 mg (2Q12) vs Ranibizumab 0.5 mg (rQ4); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Percentage Difference = -4.2, 95.1% CI 2-sided [-8.7 to 0.0] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Mean Change From Baseline in BCVA in the Study Eye at Week 52
Description: BCVA was measured using an eye chart and was reported as the number of letters read correctly using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. The study eye is defined as the eye that meets the entry criteria. If both eyes met the entry criteria, the eye with the worse BCVA at baseline (Day 1) was selected as the study eye. If both eyes had same BCVA values at baseline (Day 1), then the participant had to select their nondominant eye for treatment, or else the right eye was selected as the study eye. Mixed model for repeated measures (MMRM) analysis was used.
Time Frame: Baseline to Week 52
Population: The PP population included all randomized and treated participants without any protocol deviations that impacted the primary efficacy variable and with treatment compliance to represent the intended regimen adequately. Number of participants analyzed was based on observed data; missing data were not imputed.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Abicipar Pegol 2 mg (2Q8) | Abicipar Pegol 2 mg (2Q12) | Ranibizumab 0.5 mg (rQ4)
Number analyzed (Participants) | 241 | 239 | 272
letters | 6.7 (12.9) | 5.6 (13.3) | 8.5 (13.6)
Statistical Analysis 1: Comparison: Abicipar Pegol 2 mg (2Q8) vs Ranibizumab 0.5 mg (rQ4); Test type: Non-Inferiority — For hypothesis testing, non-inferiority of abicipar is established if the lower limit of the CI is > - 5.0 letters; Least Squares (LS) Mean Difference = -2.4, 95.1% CI 2-sided [-4.7 to -0.1], Standard Error of Mean 1.2 — MMRM included treatment, region, BL BCVA, BL CRT ≤400 or >400, choroidal neovascularization lesion type, visit, visit-by-BL BCVA interaction, and treatment-by-visit interaction term as covariates using an unstructured covariance matrix
Statistical Analysis 2: Comparison: Abicipar Pegol 2 mg (2Q12) vs Ranibizumab 0.5 mg (rQ4); Test type: Non-Inferiority — For hypothesis testing, non-inferiority of abicipar is established if the lower limit of the CI is > - 5.0 letters; LS Mean Difference = -3.7, 95.1% CI 2-sided [-6.0 to -1.3], Standard Error of Mean 1.2 — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Mean Change From Baseline in Central Retinal Thickness (CRT) in the Study Eye at Week 52
Description: CRT was assessed using spectral domain optical coherence tomography (SD-OCT), a non-invasive diagnostic system providing high-resolution imaging sections of the retina. SD-OCT was performed in the study eye after pupil dilation. A negative change from Baseline indicated improvement. The study eye is defined as the eye that meets the entry criteria. If both eyes met the entry criteria, the eye with the worse BCVA at baseline (Day 1) was selected as the study eye. If both eyes had same BCVA values at baseline (Day 1), then the participant had to select their non-dominant eye for treatment, or else the right eye was selected as the study eye. MMRM analysis was used.
Time Frame: Baseline to Week 52
Population: ITT population included all randomized participants. Number of participants analyzed was based on observed data; missing data were not imputed.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Abicipar Pegol 2 mg (2Q8) | Abicipar Pegol 2 mg (2Q12) | Ranibizumab 0.5 mg (rQ4)
Number analyzed (Participants) | 242 | 235 | 269
microns | -141.5 (136.4) | -150.1 (127.4) | -141.3 (122.0)
Statistical Analysis 1: Comparison: Abicipar Pegol 2 mg (2Q8) vs Ranibizumab 0.5 mg (rQ4); Test type: Superiority — Superiority of abicipar was demonstrated if the lower limit of CI for the treatment difference was greater than zero; LS Mean Difference = 8.6, 95.1% CI 2-sided [-3.8 to 20.9], Standard Error of Mean 6.3 — MMRM was used for analyses with covariates (treatment, region, baseline BCVA, CRT, choroidal neovascularization lesion type, visit, visit by baseline BCVA and treatment by visit interaction) with unstructured covariance matrix
Statistical Analysis 2: Comparison: Abicipar Pegol 2 mg (2Q12) vs Ranibizumab 0.5 mg (rQ4); Test type: Superiority — Superiority of abicipar was demonstrated if the lower limit of CI for the treatment difference was greater than zero; LS Mean Difference = 2.3, 95.1% CI 2-sided [-10.1 to 14.7], Standard Error of Mean 6.3 — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Percentage of Participants With a Gain of 15 or More ETDRS Letters in BCVA From Baseline in Study Eye at Week 52
Description: BCVA was measured using an eye chart and reported as the number of letters read correctly using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. The study eye is defined as the eye that meets the entry criteria. If both eyes met the entry criteria, the eye with the worse BCVA at baseline (Day 1) was selected as the study eye. If both eyes had same BCVA values at baseline (Day 1), then the participant had to select their non-dominant eye for treatment, or else the right eye was selected as the study eye.
Time Frame: Baseline to Week 52
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Abicipar Pegol 2 mg (2Q8) | Abicipar Pegol 2 mg (2Q12) | Ranibizumab 0.5 mg (rQ4)
Number analyzed (Participants) | 314 | 313 | 312
percentage of participants | 22.6 | 19.2 | 27.2
Statistical Analysis 1: Comparison: Abicipar Pegol 2 mg (2Q8) vs Ranibizumab 0.5 mg (rQ4); Test type: Superiority; Percentage Difference = -4.7, 95.1% CI 2-sided [-11.5 to 2.1] — The 95.1% CI for the weighted difference were calculated based on the Newcombe method using the Cochran-Mantel-Haenszel weights and baseline BCVA (≤55 vs >55 letters) as the stratification factor
Statistical Analysis 2: Comparison: Abicipar Pegol 2 mg (2Q12) vs Ranibizumab 0.5 mg (rQ4); Test type: Superiority; Percentage Difference = -8.2, 95.1% CI 2-sided [-14.7 to -1.5] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Mean Change From Baseline in the National Eye Institute Visual Functioning Questionnaire-25 (NEI-VFQ-25) Composite Score in Study Eye at Week 52
Description: NEI-VFQ-25 consists of 25 vision-targeted questions that represent 11 vision-related quality of life subscales and one general health item. Responses of individual participants were recorded as scores that ranged between 0 (worst) to 100 (best vision related function) with higher scale indicating better vision related function. The overall composite score is then calculated by averaging over all 11 vision-targeted subscale scores, excluding the general health score. Overall composite score was calculated based on mean of non-missing subscales. Study eye was defined as eye that meets entry criteria. If both eyes met all of entry criteria, eye with worse BCVA at baseline (day 1) was selected. If BCVA values for both eyes were identical then participant had to select non-dominant eye, or else right eye was selected as study eye. A positive change from baseline indicates improvement. MMRM analysis was used.
Time Frame: Baseline to Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Abicipar Pegol 2 mg (2Q8) | Abicipar Pegol 2 mg (2Q12) | Ranibizumab 0.5 mg (rQ4)
Number analyzed (Participants) | 250 | 253 | 273
score on a scale | 2.7 (0.7) | 3.7 (0.7) | 4.6 (0.7)
Statistical Analysis 1: Comparison: Abicipar Pegol 2 mg (2Q8) vs Ranibizumab 0.5 mg (rQ4); Test type: Superiority — Superiority of abicipar was demonstrated if the lower limit of CI for the treatment difference was greater than zero; LS Mean Difference = -1.8, 95.1% CI 2-sided [-3.7 to -0.0], Standard Error of Mean 0.9 — MMRM was used for analyses with covariates (treatment, region, baseline BCVA, visual function questionnaire (VFQ) score, visit, visit by baseline BCVA and treatment by visit interaction) with unstructured covariance matrix
Statistical Analysis 2: Comparison: Abicipar Pegol 2 mg (2Q12) vs Ranibizumab 0.5 mg (rQ4); Test type: Superiority — Superiority of abicipar was demonstrated if the lower limit of CI for the treatment difference was greater than zero; LS Mean Difference = -0.8, 95.1% CI 2-sided [-2.7 to 1.0], Standard Error of Mean 0.9 — [estimate comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: From first dose to last dose of study drug (Up to Week 104)
Description: Safety population included all treated participants.
Arm/Group | Abicipar Pegol 2 mg (2Q8) | Abicipar Pegol 2 mg (2Q12) | Ranibizumab 0.5 mg (rQ4)
All-Cause Mortality (participants affected / at risk) | 8/312 | 7/312 | 11/310
Serious Adverse Events (participants affected / at risk) | 92/312 | 102/312 | 95/310
Other Adverse Events (participants affected / at risk) | 202/312 | 217/312 | 196/310
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abicipar Pegol 2 mg (2Q8) (N=312) | Abicipar Pegol 2 mg (2Q12) (N=312) | Ranibizumab 0.5 mg (rQ4) (N=310)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 4 | 4
Coronary artery disease (Cardiac disorders) | 1 | 2 | 3
Cardiac failure congestive (Cardiac disorders) | 2 | 3 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 3 | 2
Angina pectoris (Cardiac disorders) | 0 | 1 | 2
Cardiac failure (Cardiac disorders) | 1 | 0 | 2
Arrhythmia (Cardiac disorders) | 0 | 0 | 2
Angina unstable (Cardiac disorders) | 0 | 1 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 2 | 0
Left ventricular failure (Cardiac disorders) | 1 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 1 | 0
Mitral valve prolapse (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0
Retinal artery occlusion (Eye disorders) | 1 | 3 | 1
Retinal haemorrhage (Eye disorders) | 4 | 1 | 1
Neovascular age-related macular degeneration (Eye disorders) | 0 | 1 | 1
Retinal pigment epithelial tear (Eye disorders) | 1 | 0 | 1
Macular degeneration (Eye disorders) | 0 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 1
Uveitis (Eye disorders) | 10 | 10 | 0
Iridocyclitis (Eye disorders) | 1 | 4 | 0
Retinal vasculitis (Eye disorders) | 6 | 3 | 0
Visual acuity reduced (Eye disorders) | 4 | 3 | 0
Vitritis (Eye disorders) | 5 | 2 | 0
Cataract (Eye disorders) | 3 | 1 | 0
Autoimmune uveitis (Eye disorders) | 2 | 1 | 0
Eye pain (Eye disorders) | 1 | 1 | 0
Macular fibrosis (Eye disorders) | 1 | 1 | 0
Ocular hypertension (Eye disorders) | 1 | 1 | 0
Age-related macular degeneration (Eye disorders) | 0 | 1 | 0
Iritis (Eye disorders) | 0 | 1 | 0
Macular scar (Eye disorders) | 0 | 1 | 0
Optic disc haemorrhage (Eye disorders) | 0 | 1 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 1 | 0
Vitreous adhesions (Eye disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 3 | 0 | 0
Dacryostenosis acquired (Eye disorders) | 1 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0
Necrotising retinitis (Eye disorders) | 1 | 0 | 0
Photopsia (Eye disorders) | 1 | 0 | 0
Retinal oedema (Eye disorders) | 1 | 0 | 0
Retinal tear (Eye disorders) | 1 | 0 | 0
Retinal vein occlusion (Eye disorders) | 1 | 0 | 0
Subretinal fibrosis (Eye disorders) | 1 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Femoral hernia incarcerated (Gastrointestinal disorders) | 0 | 0 | 1
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal infarction (Gastrointestinal disorders) | 0 | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 1
Death (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Asthenia (General disorders) | 1 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic mass (Hepatobiliary disorders) | 0 | 0 | 1
Biliary dilatation (Hepatobiliary disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 9 | 9 | 14
Endophthalmitis (Infections and infestations) | 1 | 4 | 2
Sepsis (Infections and infestations) | 1 | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 1 | 2
Bronchitis (Infections and infestations) | 1 | 5 | 1
Cellulitis (Infections and infestations) | 2 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1
Febrile infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 1 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 2 | 0 | 0
Abscess jaw (Infections and infestations) | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Retinitis (Infections and infestations) | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 5
Hip fracture (Injury, poisoning and procedural complications) | 1 | 3 | 3
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1 | 2
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cataract operation complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 3 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 2 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Inflammation of wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ocular procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 1
Intraocular pressure increased (Investigations) | 1 | 1 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 3 | 2
Adult failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Ankle deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 3
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bone sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastric cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Head and neck cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 2 | 5
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 2 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0
Quadrantanopia (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Dementia (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Myelopathy (Nervous system disorders) | 1 | 0 | 0
Optic neuritis (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 1
Intensive care unit delirium (Psychiatric disorders) | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1
Nephritis (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Bladder prolapse (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 2 | 2
Aortic stenosis (Vascular disorders) | 0 | 2 | 1
Hypertension (Vascular disorders) | 2 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abicipar Pegol 2 mg (2Q8) (N=312) | Abicipar Pegol 2 mg (2Q12) (N=312) | Ranibizumab 0.5 mg (rQ4) (N=310)
Conjunctival haemorrhage (Eye disorders) | 27 | 32 | 46
Neovascular age-related macular degeneration (Eye disorders) | 26 | 28 | 39
Eye pain (Eye disorders) | 26 | 26 | 22
Cataract (Eye disorders) | 29 | 19 | 20
Visual acuity reduced (Eye disorders) | 24 | 33 | 18
Vitreous detachment (Eye disorders) | 19 | 21 | 17
Retinal haemorrhage (Eye disorders) | 16 | 23 | 16
Vitreous floaters (Eye disorders) | 22 | 20 | 16
Eye irritation (Eye disorders) | 11 | 16 | 9
Subretinal fluid (Eye disorders) | 8 | 17 | 7
Iridocyclitis (Eye disorders) | 10 | 18 | 2
Nasopharyngitis (Infections and infestations) | 37 | 36 | 36
Urinary tract infection (Infections and infestations) | 19 | 21 | 31
Influenza (Infections and infestations) | 15 | 16 | 24
Bronchitis (Infections and infestations) | 23 | 19 | 23
Conjunctivitis (Infections and infestations) | 21 | 20 | 11
Fall (Injury, poisoning and procedural complications) | 11 | 12 | 17
Intraocular pressure increased (Investigations) | 15 | 25 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 21 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 18 | 10
Hypertension (Vascular disorders) | 25 | 20 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT02462928/SAP_000.pdf
  • Study Protocol (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT02462928/Prot_001.pdf